CLINICAL TRIAL: NCT04489953
Title: Optimizing Antiretroviral Treatment Switch in HIV-Infected Ugandan Children
Brief Title: Comparison of Treatment Failure Criteria in HIV-Infected Children in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MU-JHU CARE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9415
Record Dates: First submitted 2020-07-13; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: HIV
MeSH Terms: interventions — Viral Load

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical and Immunologic criteria (Active Comparator): In the clinical and immunologic monitoring criteria was based on the 2010 WHO guidelines. Whereby children were monitored using clinical presentation and CD4 count to define treatment failure.
  Interventions: Other: Viral Load
- Clinical, Immunologic and Virologic criteria (Active Comparator): In the Clinical, Immunologic and Virologic criteria was based on a confirmed viral load of > 1000 HIV RNA copies/ml; as well as clinical and immunologic criteria
  Interventions: Other: Viral Load

INTERVENTIONS:
Other: Viral Load — For the Clinical and Immunologic criteria, viral load was done retrospectively on stored plasma samples. Whereas for the Clinical, Immunologic and Virologic criteria, viral load was done in real-time

SUMMARY:
The main goal was to compare clinical and immunological versus clinical, immunological plus viral load criteria for switching to second-line ART by comparing 48 week treatment outcomes, including survival rates, viral suppression, failure to thrive, and AIDS-defining illnesses for treatment experienced children randomized to two switching criteria.

DETAILED DESCRIPTION:
The overall goal of the study was aimed at determining whether the use of the current WHO criteria alone (clinical and immunologic) to define treatment failure as the trigger for switching to second-line antiretroviral therapy leads to poorer 6 month and 12 month treatment outcomes when compared to combining clinical and immunologic parameters with viral load (VL) monitoring.

In addition the study aimed at obtaining plasma samples from treatment experienced children, for future resistance testing. The results of this study may help guide WHO and national pediatric ART programs on the need for routine VL monitoring for children initiating HAART in resource limited settings, where virologic tests including resistance testing are not readily available or affordable.

ELIGIBILITY:
Inclusion Criteria:

* HIV-Infected Children, 1 year to 12 years
* ART experienced and enrolled in an existing treatment program that used clinical and immunologic criteria to monitor response to ART.

Exclusion Criteria:

* None

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Criteria for switching HIV-Infected Children to second line | 2 years
  Confirmed viral load > 1,000 HIV RNA copies/ml

REFERENCES:
- [Derived] Kibalama Ssemambo P, Nalubega-Mboowa MG, Owora A, Serunjogi R, Kironde S, Nakabuye S, Ssozi F, Nannyonga M, Musoke P, Barlow-Mosha L. Virologic response of treatment experienced HIV-infected Ugandan children and adolescents on NNRTI based first-line regimen, previously monitored without viral load. BMC Pediatr. 2021 Mar 22;21(1):139. doi: 10.1186/s12887-021-02608-0. PMID 33752636